CLINICAL TRIAL: NCT05145790
Title: State of Play in Strasbourg University Hospital of the Place of Consultations Specializing in the Diagnosis of Mood Disorders
Brief Title: The Place of Consultations Specializing in the Diagnosis of Mood Disorders in Strasbourg University Hospital
Acronym: MOOD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8365
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Mood Disorders
Keywords: Mood Disorders
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mood disorders (depressive disorders and bipolar disorders) are among the ten most worrying diseases of the 21st century according to the WHO.

In order to support psychiatrists in their diagnostic reflection, structures have been created. Since 2009, the Psychiatry Service 2 within the Psychiatry, Mental Health and Addictology Pole of the University Hospitals of Strasbourg has offered specialized consultations in mood disorders.

More than 10 years after the creation of these consultations, it seems interesting to study the profile of the users and to describe the nature of the reports of these in-depth evaluation consultations (diagnosis, therapeutic advice)

ELIGIBILITY:
Inclusion criteria:

* Major subject
* Specialized primary consultation highlighting symptoms of mood disorders with Prof. Berstchy in the psychiatry department 2 in the University Hospital of Strasbourg (patients whose consultation request was linked to symptoms or a diagnosis of ADHD will not be included in the study population).
* Consultation that took place in 2018 and 2019.
* Patient who did not express his opposition to the reuse of his data for scientific research purposes.

Exclusion criteria:

* Patient opposition to the use of their personal data for scientific research purposes.
* Prior existence of a previous specialist consultation in mood disorders with Prof. Berstchy (the information collected during the first consultation is not accessible)
* Patient under curatorship, guardianship or legal protection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject with pecialized primary consultation highlighting symptoms of mood disorders
Sampling Method: Non-Probability Sample
Enrollment: 197 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Descriptive study of the clinical characteristics of patients coming to consultations specializing in mood disorders in Strasbourg University Hospitals | Files analysed retrospectively from January 01, 2018 to December 31, 2019 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Gilles BERTSCHY, MD, PhD, Principal Investigator — Service de psychiatrie 2 - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de psychiatrie 2 - Hôpitaux Universitaires de Strasbourg, Strasbourg, France